CLINICAL TRIAL: NCT01242995
Title: Prospective Evaluation of the Clinical Utility of the Thin Scope/Anchoring Balloon Cholangiopancreatoscopy System for Disorders fo the Pancreatobiliary System
Brief Title: Endoscopic Retrograde Cholangiopancreatography (ERCP) With Cholangiopancreatoscopy Using a Thin Scope
Status: Withdrawn | Type: Observational
Why Stopped: The device was withdrawn from clinical use
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Thin Scope
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Disorders of the Pancreatobiliary System
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pancreatobiliary disorders/thin scope: All patients will be evaluated with cholangioscopy and/or pancreatoscopy using the thin scope.
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP)with Cholangiopancreatoscopy using the thin scope

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP)with Cholangiopancreatoscopy using the thin scope — Endoscopic Retrograde Cholangiopancreatography (ERCP) with cholangiopancreatoscopy using the thin scope system.

SUMMARY:
The purpose of this study is to evaluate the use of a thin scope/anchoring Balloon endoscopy system for the medical care of pancreatic and/or biliary disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subject has clinical indication for Endoscopic Retrograde Cholangiopancreatography (ERCP) with Cholangioscopy and/or pancreatoscopy
3. Subject must be able to give informed consent.

Exclusion Criteria:

1. Any contraindication to Endoscopic Retrograde Cholangiopancreatography (ERCP)
2. The subject is unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a medical indication for Endoscopic Retrograde Cholangiopancreatography (ERCP) with cholangioscopy and/or pancreatoscopy and are referred for the procedure as part of their standard medical care will be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
use of a thin endoscope system for the evaluation and/or treatment of pancreatobiliary disorders. | approxiamtely 2-4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter Draganov, MD, Principal Investigator — University of Florida